CLINICAL TRIAL: NCT01594346
Title: Multicenter Vitamin E Trial in Aging Persons With Down Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Institute for Basic Research (Other Government)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); New York State Psychiatric Institute (Other); University of California, San Diego (Other); Columbia University (Other); Bronx Veterans Medical Research Foundation, Inc (Other)
Responsible Party: Principal Investigator, Arthur Dalton, Deputy Director, New York State Institute for Basic Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCT00056329; R01AG016381 (NIH)
Record Dates: First submitted 2012-05-02; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease; Down Syndrome
Keywords: Vitamin E; alpha-tocopherol; cognitive decline; Down syndrome; Aging; Dementia
MeSH Terms: conditions — Alzheimer Disease; Down Syndrome; Cognitive Dysfunction; Dementia | interventions — alpha-Tocopherol; Vitamin E; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill
- Alpha-Tocopherol (Active Comparator)
  Interventions: Drug: Alpha-Tocopherol

INTERVENTIONS:
Drug: Alpha-Tocopherol — 1,000 International Units, two times a day for 36 months
  Other Names: Vitamin E
  Arms: Alpha-Tocopherol
Drug: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of 2,000 international units of Vitamin E (alpha tocopherol)on cognitive function of aging persons with Down syndrome. It is a randomized, double-blind, placebo-controlled trial lasting 36 months. It is expected that Vitamin E will slow the deterioration in cognitive functions associated with Alzheimer disease.

DETAILED DESCRIPTION:
Alzheimer disease (AD) continues to be the most serious health problem faced by aging persons with Down syndrome. AD is also a major public health concern in the aging general population. With increasing life expectancy there will be a dramatic increase in the prevalence of AD cases, which will pose a significant increased burden on the health care system and individual providers of care. Persons with Down syndrome are uniquely vulnerable to a form of Alzheimer disease indistinguishable from the sporadic variety that affects aging individuals from the general population. Oxidative damage is a highly plausible mechanism in the pathogenesis of this disease due to the overexpression of superoxide dismutase, associated with a gene located on chromosome 21, which is present in triplicate in the Down syndrome genotype. For the last six years, we have been conducting a clinical trial to determine the safety and efficacy of the anti-oxidant Vitamin E in slowing the cognitive and functional decline associated with the dementia of AD among individuals with DS. The study is a randomized, double-blind trial, stratified in a two-arm parallel design. The subjects are medically stable individuals who are 50 years of age or older at the time of screening. Among those randomized to the treatment arm, vitamin E is taken in the form of 1000 IU capsules for 36 months. Each subject is evaluated every 6 months for 3 years. The primary outcome is is the Brief Praxis Test (BPT), which is well-suited to quantifying cognitive decline in this population. The target enrollment of 350 persons is estimated to be sufficient to provide adequate statistical power to detect a slowing by one-third in the rate of cognitive decline with vitamin E treatment. The Data and Safety Monitoring Board (DSMB) for this trial includes 4 physicians, and a statistician with expertise in clinical trials. Each DSMB member receives a report on each serious adverse event (SAE) on a flow basis, and statistically summaries of unblinded safety data--including deaths, adverse events and vital signs--prior to each meeting of the DSMB. The most recent DSMB meeting took place on February 23,2010. The timeline for study completion is: recruitment of the study sample (N=350) was completed on 12/31/2008; the final 36-month evaluation will take place in 04/2010; statistical analysis and final report of results is expected to be completed by 12/31/2010.

ELIGIBILITY:
Inclusion Criteria:

* presence of clinically determined Down syndrome (karyotypes optional)
* appropriately signed and witnessed consent form
* age of 50 years or older at the start of the protocol
* medically stable
* medications stable more than 1 month
* involvement/cooperation of informant/caregiver

Exclusion Criteria:

* medical/neurological condition (other than Alzheimer disease) associated with dementia
* inability to adequately perform the Brief Praxis Test, as demonstrated by a score <20
* in the presence of dementia, modified Hachinski score > 4 at Screening Visit
* major depression within 3 months
* history of coagulopathy (inherited or acquired)
* current use of anticoagulants
* use of experimental medications within 2 months
* regular use of vitamin E greater than 50 units per day during the previous 6 months
* allergy to vitamin E

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2000-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The Brief Praxis Test | 36 months

SECONDARY OUTCOMES:
The Fuld Object Memory Test | 36 Months
New Dot Test | 36 Months
Orientation Test | 36 Months
Vocabulary Test | 36 Months
Behavior and Function | 36 Months
Clinical Global Impression | 36 Months
Incident Dementia | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Aisen, M.D., Study Director — University of California, San Diego; Mary C. Sano, Ph.D., Study Director — Bronx Veterans Medical Research Foundation; Howard F. Andrews, Ph.D., Study Director — New York Psychiatric Institute; Wei-Yann Tsai, Ph.D., Study Director — Columbia University